CLINICAL TRIAL: NCT04568265
Title: A Multicenter, Open-label, Phase II Clinical Study to Evaluate the Safety and Efficacy of APG-1387 in Combination With Entecavir in Patients With Chronic Hepatitis B
Brief Title: A Clinical Study of APG-1387 in Combination With Entecavir in Patients With Chronic Hepatitis B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascentage Pharma Group Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APG1387BC201
Record Dates: First submitted 2020-09-24; First posted 2020-09-29 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Hepatitis B; Chronic Hep B; HBV
Keywords: HBeAg-positive; HBeAg-negative
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — APG-1387; entecavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- APG-1387 12 mg combined with entecavir 0.5 mg (Experimental)
  Interventions: Drug: APG-1387; Drug: Entecavir 0.5 mg
- APG-1387 20 mg combined with entecavir 0.5 mg (Experimental)
  Interventions: Drug: APG-1387; Drug: Entecavir 0.5 mg
- APG-1387 30 mg combined with entecavir 0.5 mg (Experimental)
  Interventions: Drug: APG-1387; Drug: Entecavir 0.5 mg
- entecavir 0.5 mg (Experimental)
  Interventions: Drug: Entecavir 0.5 mg

INTERVENTIONS:
Drug: APG-1387 — Weekly intravenous infusion for 30 minutes
  Arms: APG-1387 12 mg combined with entecavir 0.5 mg; APG-1387 20 mg combined with entecavir 0.5 mg; APG-1387 30 mg combined with entecavir 0.5 mg
Drug: Entecavir 0.5 mg — Taken daily by mouth
  Other Names: Baraclude

SUMMARY:
This study is a multicenter, open-label, phase II clinical study in subjects with chronic hepatitis B (CHB), to characterize the safety, tolerability, pharmacokinetic profile and preliminary anti-hepatitis B virus (HBV) efficacy of APG-1387 in combination with entecavir, and to determine the optimal dose of APG-1387 in combination with entecavir.

DETAILED DESCRIPTION:
The study is divided into two parts:

Part 1 will evaluate the safety, tolerability, and pharmacokinetics of APG-1387 in combination with entecavir, including determination of the maximum tolerated dose (MTD)/ recommended dose in patients with CHB. APG-1387 will be administered once weekly via intravenous infusion for 30 minutes for consecutive 4 weeks. APG-1387 will be escalated at 3 dose cohorts of 12 mg, 20 mg, and 30 mg. Entecavir will be administered orally at 0.5 mg daily for 12 weeks: in combination with APG-1387 for the first 4 weeks, followed by entecavir maintenance monotherapy for additional 8 weeks. The total treatment duration will be 12 weeks.

Part 2 is a randomized, parallel, open-label study to investigate the preliminary anti-HBV efficacy of APG-1387 in combination with entecavir compared with entecavir monotherapy. CHB subjects will be randomly assigned to one of 4 cohorts at 1:1:1:1, including APG-1387 at 3 different doses (12 mg, 20 mg, and 30 mg) in combination with entecavir for 12 weeks, respectively, then continued entecavir monotherapy for additional 12 weeks; and one entecavir monotherapy cohort for 24 weeks. The course of treatment is 24 weeks in all cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) within the range of 18 - 27.9
* Documented chronic HBV infection (e.g., HBsAg positive for at least 6 months).
* HBeAg-positive or HBeAg-negative
* Treatment-naïve and treatment-experienced subjects are required to:

  1. Treatment-naïve subjects:

     * No antiviral therapies including nucleos(t)ide analogues or immunomodulators such as interferon within 180 days prior to screening
     * HBV DNA ≥ 2x10˄3 IU/mL for HBeAg negative subjects and ≥ 2x10˄4 IU/mL for HBeAg positive subjects (PCR)
     * Alanine transaminase (ALT) ≥ upper limit of normal (ULN) and < 10 × ULN (and excluding ALT elevation caused by non-HBV reasons such as drug or alcohol consumption)
  2. Treatment-experienced subjects:

     * Using entecavir > 180 days prior to screening, and should continue the treatment regimen until enrolled into the study
     * HBV DNA less than the lower limit of quantification (LLOQ) or < 20 IU/mL (PCR)
     * ALT < 1.5 × ULN
* Adequate hematological function:

  * White blood cell count (WBC) ≥ 3.5 × 10˄9/L
  * Hemoglobin ≥ 120 g/L for males and ≥ 110 g/L for females
  * Platelet count ≥ 100 × 10˄9/L
* Adequate renal and liver function:

  * Serum creatinine ≤ 1×ULN
  * Serum albumin ≥ 35.0g/L
  * Urine protein is negative or 1 + (re-examination is required when 1 + or 24-hour urine protein quantification is added when necessary. If it turns negative or is within the normal range, it can be included)
  * Estimated creatinine clearance (CLCr) ≥ 50 mL/min based on serum creatinine measured at the screening assessment and actual body weight (calculated creatinine clearance by the Cockcroft-Gault formula)
  * Total bilirubin ≤1.5×ULN
  * International normalized ratio (INR) ≤ 1.5×ULN
  * Alkaline phosphatase ≤ 2.5×ULN
* Female subjects of childbearing potential should have a negative serum pregnancy test within 7 days prior to the first dose
* Subjects and theirs partners are willing to use effective contraception as defined in the protocol during the treatment and for at least 6 months after the last dose of study drug
* Ability to understand and willingness to sign a written informed consent form (the consent form must be signed by the subject prior to any study-specific procedures)
* Willingness and ability to comply with study procedures and follow-up examination

Exclusion Criteria:

* Co-infection with HIV, hepatitis C virus (HCV), or hepatitis delta virus (HDV); or other active and severe infections
* Syphilis with positive antibody for treponema pallidum
* Subjects with liver disease other than hepatitis B, including but not limited to chronic alcoholic hepatitis, drug-induced liver injury, autoimmune liver disease, hereditary liver disease (such as Wilson's disease), and active hepatitis due to other causes
* History or manifestation of hepatic decompensation (e.g., Child-Pugh Class B or C, or history of ascites, gastrointestinal bleeding, hepatic encephalopathy, or spontaneous bacterial peritonitis)
* Progressive fibrosis/cirrhosis, defined by liver fibrosis scan ≥ 12 kilopascal (kPa) at screening, or cirrhosis diagnosed by imaging examinations, or Metavir score F3, F4 fibrosis on liver biopsy at any time
* Clinically diagnosed hepatocellular carcinoma, or diagnosis of hepatocellular carcinoma cannot be excluded, or serum alpha-fetoprotein greater than 50 μg/L
* History of malignancy (except cured and no evidence of recurrence of basal cell carcinoma of the skin or situ cervical cancer) or lymphoproliferative disease
* History of neurological or mental disorders, such as epilepsy, dementia, and poor compliance
* Uncontrolled primary diseases of other important organs, such as clear medical history of nervous system, cardiovascular system, urinary system (including chronic or intermittent urinary system diseases), digestive system, respiratory system, endocrine/metabolic and musculoskeletal system, such as poorly controlled diabetes, hypertension, etc., making the investigator consider the subject unsuitable
* QTcB [QTcB = QT/(RR^ 0.5); RR is the normalized heart rate value, obtained by dividing 60 by heart rate in seconds; other parameters in milliseconds] > 450 milliseconds for men and > 470 milliseconds for women; any clinically important abnormality in the rhythm, conduction, or morphology of the resting electrocardiogram (ECG) (e.g., complete left bundle branch block, third degree heart block, second degree heart block); congenital long QT syndrome or family history of long QT syndrome
* History of alcoholism (mean daily intake of ethanol ≥ 30 g (male) or ≥ 20 g (female) within 1 year), and drug abuse
* Subjects planning to become pregnant within 1 year, who are pregnant or breastfeeding
* Received or may receive continuous treatment with immunomodulators (e.g., steroids) or biological agents (e.g., monoclonal antibodies, interferons) within 3 months before screening
* Participated in clinical trials within 3 months before screening
* Trauma or major surgical operation within 4 weeks before screening
* Previous treatment with inhibitors of apoptosis proteins
* Any subject considered unsuitable for the trial by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) rate at each dose level | 28 days
  DLT will be assessed within the first 28-day cycle of study treatment via NCI CTCAE version 5.0
Decline in Hepatitis B surface Antigen (HBsAg) | 12 weeks
  The difference in HBsAg decline between APG-1387 combined with entecavir arms and entecavir monotherapy arm

CONTACTS AND LOCATIONS:
Overall Officials: Yifan Zhai, MD, PhD, Study Chair — Ascentage Pharma Group Inc.
Locations (4):
- China (4):
  - Guangzhou Eighth People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No